CLINICAL TRIAL: NCT07234825
Title: Trial of Partial Enteral Nutrition With Dairy Free Diet in Eosinophilic Esophagitis Induction of Remission
Brief Title: Trial of Partial Enteral Nutrition With Dairy Free Diet in Eosinophilic Esophagitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kate Farms Inc (Industry)
Collaborators: Seattle Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Seattle2025
Record Dates: First submitted 2025-11-13; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Eosinophilic Esophagitis (EoE)
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — penclomedine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): 12 participants will be control subjects without diagnosis of EoE
- Dairy Free (Experimental): 12 subjects will be enrolled in the dairy free diet group.
  Interventions: Other: Dairy elimination alone
- Dairy free + Partial Enteral Nutrition (PEN) diet (Experimental): 12 subjects will be enrolled in the diary free and 50% PEN diet
  Interventions: Other: Partial enteral nutrition (PEN) with dairy elimination

INTERVENTIONS:
Other: Partial enteral nutrition (PEN) with dairy elimination — Patients in the PEN with dairy elimination group will receive 50% calories from Kate Farms Standard 1.2 formula and 50% dairy free regular diet.
  Arms: Dairy free + Partial Enteral Nutrition (PEN) diet
Other: Dairy elimination alone — Participants in this group will be on a dairy-free regular diet alone.
  Arms: Dairy Free

SUMMARY:
This study aims to introduce a new dietary therapy for Eosinophilic Esophagitis (EoE) patients by using partial enteral nutrition (PEN) to enhance remission rates and explore how this approach affects immune function, gut microbiota, and environmental toxin exposures.

DETAILED DESCRIPTION:
The purpose of this research project is to offer patients diagnosed with Eosinophilic Esophagitis (EoE) a novel dietary therapy approach which models that of evidence-based dietary therapy used in Crohn's disease and the principles of dietary antigen elimination currently successfully implemented in EoE patients. The study proposes using partial enteral nutrition (PEN) to improve remission rates in EoE patients and investigate the mechanism by which these effects immune dysregulation, microbiota shifts, and through assessment of changes in environmental toxin exposure.

Objectives 1: Determine clinical and endoscopic remission rates, adherence, nutrition, and anthropometric measures in EoE patients prior to and three months after PEN with dairy elimination.

Objectives 2: Investigate immune profiles in EoE patients prior to and three months after PEN with dairy elimination.

Objectives 3: Investigate the microbiota in EoE patients prior to and three months after PEN with dairy elimination.

Objectives 4: Investigate environmental contaminants prior to and three months after PEN with dairy elimination.

It is hypothesized favorable shifts in the microbiota, immune system, and environmental contaminants will be present following three months of PEN in the EoE patient population.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients 1 year to 21 of age presenting with chronic symptoms of dysphagia, odynophagia, vomiting or heartburn, chronic abdominal pain, weight loss, picky eating, to outpatient gastroenterology clinic and are planning to undergo EGD for evaluation.

Exclusion Criteria:

* Non-English-Speaking Subjects, adults unable to consent, wards of the state, pregnant women, and prisoners will be excluded from the study.
* Patients with autoimmune conditions such as inflammatory bowel disease. Patients with prior esophageal or intestinal surgeries.
* Patients with history of eating disorders or ARFID.
* Patients with fistulizing or fibrotic disease on baseline EGD.
* Patients who have received proton pump inhibitory therapy in the past month.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of PEN assessed by 3-day diet record | 3 months
  Feasibility and adherence of PEN in EoE patients will be evaluated using 3-day diet records collected at 2 weeks post initiation of the study and at 3 months.
Tolerability of PEN in EoE patients will be assessed by stool quality evaluated using the Bristol Stool Chart. | 3 months
  Bristol stool chart will be used to assess stool quality at 2 weeks and at month 3.
Clinical and endoscopic remission rates assessed by mucosal eosinophilia and Eosinophilic Esophagitis Histology Scoring System (EoE-HSS) from GI tissue biopsies | 3 months
  For baseline and three-month tissue collection, GI tissue biopsies will be obtained at the time of clinical endoscopy assess mucosal eosinophilia and EoE-HSS.
Immune profiles assessed by blood markers | 3 months
  Immune profiles in EoE patients will be assessed by blood markers using CBC with differential, comprehensive metabolic panel, C-Reactive Protein, and Erythrocyte Sedimentation Rate before and after PEN and dairy elimination.
Microbiota shifts in EoE patients | 3 months
  Microbiota shifts will be assessed from stool metabolomics, urine metabolomics, oral swab microbiome, and esophageal brushing of EoE before and after PEN and dairy free diets.
Environmental contaminants assessed by blood serum levels | 3 months
  Environmental contaminants assessed by CBC with differential before and after PEN with dairy elimination.

SECONDARY OUTCOMES:
Nutritional status assessed by 3-day diet record and blood collection | 3 months
  Nutrition status of EoE will be assessed by the collection a 3-day diet record, vitamin D, vitamin B12, iron, total iron binding capacity, and ferritin at baseline and 3 months.
Growth and development assessed by anthropometric measure | 3 months
  Z-scores for height and weight will be collected at baseline and at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pickens, DO, Principal Investigator — Seattle Children's Hospital

IPD SHARING:
Plan to Share IPD: No